CLINICAL TRIAL: NCT03683485
Title: Long-duration (3 Minutes) Endoscopic Papillary Balloon Dilation Versus Endoscopic Sphincterotomy in Patients With a Naive Major Papilla and Small- to Medium Sized Biliary Stones: Multicenter, Randomized, Controlled Trial
Brief Title: Long-duration EPBD vs EST for Removal of Biliary Stones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dankook University (Other)
Collaborators: Inje University (Other); The Catholic University of Korea (Other); Wonkwang University (Other)
Responsible Party: Principal Investigator, Jun Ho Choi, Assistant Professor, Dankook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-03-009
Record Dates: First submitted 2018-04-05; First posted 2018-09-25 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Cholangiopancreatography, Endoscopic Retrograde
Keywords: Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- long duration EPBD group (Experimental): Balloon dilation was performed using wire-guided hydrostatic balloon catheters. An 8-mm dilatation balloon was used for EPBD. Balloons were gradually inflated to maximum pressure for 3 minute, and complete inflation was verified by fluoroscopy. Stones were removed by standard techniques, including balloon or basket catheters.
  Interventions: Procedure: long duration EPBD; Procedure: EST
- endoscopic sphincterotomy (EST) group (Active Comparator): After deep cannulation was achieved, a complete sphincterotomy was performed with a 25-mm pull-type sphincterotome (Clever Cut 3; KD-V411M, Olympus, Tokyo, Japan) and the sphincter was divided up to the transverse duodenal fold. A complete sphincterotomy was defined by the free passage of a fully bowed sphincterotome and the presence of spontaneous bile drainage. A complete sphincterotomy was defined by the free passage of a fully bowed sphincterotome and the presence of spontaneous bile drainage.
  Interventions: Procedure: long duration EPBD; Procedure: EST

INTERVENTIONS:
Procedure: long duration EPBD — An 8-mm dilatation balloon was used for EPBD. Balloons were gradually inflated to maximum pressure for 3 minute, and complete inflation was verified by fluoroscopy.
Procedure: EST — After deep cannulation was achieved, a complete sphincterotomy was performed with a 25-mm pull-type sphincterotome (Clever Cut 3; KD-V411M, Olympus, Tokyo, Japan) and the sphincter was divided up to the transverse duodenal fold.

SUMMARY:
Although EPBD has a lower risk of post-ERCP bleeding and long-term complications than EST and is easier to perform in altered/difficult anatomy, EPBD is reserved for patients with bleeding diathesis by current consensus because some studies reported a higher risk of pancreatitis. However, recent meta-analyses indicate that short EPBD duration increases the risk of post-ERCP pancreatitis, and EPBD with adequate duration has a similar pancreatitis risk and a lower overall complication rate compared with EST for choledocholithiasis.

Therefore, this study aim to compare long-duration EPBD vs EST in the treatment of extrahepatic biliary stones.

DETAILED DESCRIPTION:
Gallstones occur in 10%-15% of adults in the United States and are the most common and costly digestive disorder. Concomitant bile duct stones occur in up to 15% of persons with symptomatic gallstones. Endoscopic retrograde cholangiopancreatography (ERCP) with sphincterotomy is the standard treatment for removal choledocholithiasis. The biliary sphincter is permanently ablated by sphincterotomy. Enteric-biliary reflux occurs with bacterial colonization, increased bile lithogenicity, contamination with cytotoxins, and chronic inflammation of the biliary system. Endoscopic papillary balloon dilation (EPBD) has become an option for removal of stones 1 cm or smaller in size. Advantages of EPBD over EST include a decreased risk of post-ERCP bleeding as well as a decreased risk of stone recurrence and cholangitis. Although a short dilation duration (≤1 minute) was previously advocated, a study that performed EPBD for 1 minute observed a 15.4% risk of post-ERCP pancreatitis with 2 cases of mortality. European Society of Gastrointestinal Endoscopy guideline recommends that the duration of EPBD should exceed 2 minutes because long-duration EPBD (>1 minute) is preferred over short-duration EPBD (≤1 minute) with better outcomes. A meta-analysis of RCTs showed that the duration of EPBD is inversely associated with the risk of PEP. Previous RCTs comparing outcome between EPBD and EST used short EPBD duration between 25 seconds and 1 minute, and there has been no comparison of outcome between EST and long-duration EPBD. The aim of this study was to compare the early and long term outcomes of patients treated with long duration balloon dilation or sphincterotomy for extraction of bile duct stones in a randomized, multicenter fashion involving a broad spectrum of practices.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients were invited to participate by the investigators or research staff if they were at least 18 years old,
* patients who had known or suspected choledocholithiasis

Exclusion Criteria:

* active acute pancreatitis
* septic shock,
* coagulopathy (international normalized ratio >1.2, partial thromboplastic time greater than twice that of control),
* platelet count <50,000 x 103/uL,
* anticoagulation therapy within 48 hours of the procedure,
* stone diameter > 8 mm,
* bile duct diameter >15 mm, prior sphincterotomy,
* need for precut sphincterotomy for biliary access,
* biliary stricture,
* Billroth II or Roux-en-Y anatomy,
* periampullary malignancies,
* primary sclerosing cholangitis, pregnancy,
* and inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
rate of adverse event | up to 1 month after ERCP
  Number of participants with treatment-related adverse events

SECONDARY OUTCOMES:
the stone clearance rate at the index ERCP | during ERCP
  complete extraction of choledocholithiasis of all stones, fragments, and sludge at the initial procedure
direct cost | within 30 day after ERCP
  The direct cost included the total cost for the entire admission, which comprised costs of hospital stay, performed procedures, and management of complications
recurrence of choledocholithiasis | more than 3 year follow-up
  recurrent choledocholithiasis or acute cholangitis either with or without bile duct stones, and overall hepatobiliary complications
adverse event (pancreatitis) | up to 1 month after ERCP
  rate of pancreatitis
adverse event (bleeding) | up to 1 month after ERCP
  rate of bleeding
adverse event (cholangitis) | up to 1 month after ERCP
  rate of cholangitis

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ho Choi, MD, PhD, Principal Investigator — Dankook University
Locations (4):
- South Korea (4):
  - Dankook University College of Medicine, Cheonan, Chungcheongnam-do
  - Wonkwang University, Iksan, Jeollabukdo
  - Inje University, Haeundae Paik Hospital, Busan
  - St. Mary's Hospital, The Catholic University of Korea,, Daejeon